CLINICAL TRIAL: NCT01320709
Title: Single-center, Randomized, Placebo-controlled, Double-blind, Parallel Group Study to Evaluate Whether a Single-dose of Either 20 mg Piroxicam, 40 mg Piroxicam or 80 mg Piroxicam Shows an Effect on Ovulation After the Onset of LH Surge Compared to Placebo in Healthy Young Women
Brief Title: Effect of Piroxicam on Ovulation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 14835; 2010-021195-28 (EudraCT Number)
Record Dates: First submitted 2011-03-21; First posted 2011-03-22 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2014-12

CONDITIONS: Contraception, Postcoital
Keywords: Emergency contraception; Contraception
MeSH Terms: interventions — Piroxicam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Experimental)
  Interventions: Drug: Piroxicam ( BAYl1902)
- Arm 2 (Experimental)
  Interventions: Drug: Piroxicam ( BAYl1902)
- Arm 3 (Placebo Comparator)
  Interventions: Drug: Placebo
- Arm 4 (Experimental)
  Interventions: Drug: Piroxicam ( BAYl1902)

INTERVENTIONS:
Drug: Piroxicam ( BAYl1902) — Single dose of 20 mg piroxicam (i.e., 1 piroxicam capsule + 3 placebo capsule)
  Arms: Arm 1
Drug: Piroxicam ( BAYl1902) — Single dose of 40 mg piroxicam (i.e., 2 piroxicam capsules + 2 placebo capsule)
  Arms: Arm 2
Drug: Placebo — Single dose of placebo (i.e., 4 placebo capsules)
  Arms: Arm 3
Drug: Piroxicam ( BAYl1902) — Single dose of 80 mg piroxicam (i.e., 4 piroxicam capsules)
  Arms: Arm 4

SUMMARY:
In this study the effect of piroxicam on the ovulation will be evaluated. Therefore piroxicam will be administered as a single-dose after onset of LH surge (luteinizing hormone, hormone which triggers ovulation).

Additionally blood levels of endogenous hormones (hormones produced by your body) will be measured and transvaginal ultrasound examinations will be conducted at regular intervals. In addition the concentration of piroxicam in blood will be determined in regular intervals.

With regards to the tolerability of the study drug subjects will be asked regularly how they feel.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent available before any study specific tests or procedures are performed
* Healthy female subject
* Age: 18 to 35 years (inclusive) at the first screening visit
* Body mass index (BMI ): 18-30 kg/m² (inclusive) at the first screening visit
* Confirmation of the subject's health insurance coverage prior to the first screening visit
* Willingness to use non-hormonal methods of contraception during the study
* Ability to understand and follow study-related instructions
* Adequate venous access

Exclusion Criteria:

* Incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination, and effects of the study drugs will not be normal
* Hypersensitivity to the active substance or skin reactions (irrespective of severity) to piroxicam, non-steroidal anti-inflammatory drugs or other medicinal products in the past
* History or presence of inflammatory diseases of the gastrointestinal tract, gastrointestinal bleeding, ulcers or perforation
* Regular intake of medication other than hormonal contraceptives
* Clinically relevant findings in the gynecological examination including transvaginal ultrasound (TVU)
* Clinically relevant findings in the physical examination, especially signs of bleeding diathesis or heart failure
* Time point "onset of LH surge" in the pre-treatment cycle not determinable
* Time point "ovulation" in the pre-treatment cycle not determinable
* Lacking suitability for frequent TVU examinations
* History or presence of suffering from hay fever

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2011-03; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Effect of piroxicam on ovulation (delay or inhibition) when given after the onset of LH surge | after 2 months

SECONDARY OUTCOMES:
course of follicle sizes | after 2 months
course of gonadotropins (follicle-stimulating hormone [FSH], LH) and ovarian steroids (estradiol [E2], progesterone) | after 2 months
Concentration-times courses of piroxicam | after 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Berlin, State of Berlin, Germany